CLINICAL TRIAL: NCT07359716
Title: Virtual Reality Verses Conventional Physical Therapy in Parkinson's Disease Patients
Acronym: VR-CPT-PD Stud
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montiha Azeem (Other)
Responsible Party: Sponsor-Investigator, Montiha Azeem, Principal investigator, University of Lahore
Organization: University of Lahore (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC-UOL-/342/08/24
Record Dates: First submitted 2026-01-01; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Parkinson s Disease
Keywords: parkinson's disease; virtual reality rehabilitation; conventional physical therapy; balance training
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A Conventional physical therapy (Experimental): The goal is to target the domains of balance and gait through interactive virtual reality-based tasks that provide real-time feedback and motivational engagement. Equipment will include either immersive or semi-immersive virtual reality systems or balance-platform-based exergames, with motion sensors or inertial measurement units to capture movements. Safety harnesses or gait belts will be used where required. The session will begin with the 5-minute warm-up as the cpt group. Fifteen minutes of virtual reality balance modules will include weight-shifting games, stepping to virtual targets, sensory manipulation with altered virtual environments, and real-time feedback through visual and auditory cues. Difficulty will be progressed by increasing speed, accuracy demands, or reducing time allowances. This will be followed by 10-12 minutes of virtual reality gait and dynamic tasks, such as treadmill walking with augmented environments, step length and cadence targets, and obstacle avoidanc
  Interventions: Behavioral: Conventional Physical Therapy
- group B Virtual Reality-Based Physical Therapy (Experimental): The objective is to improve dynamic balance, gait, mobility, and reduce fall risk using evidence-based conventional approaches. Each session will begin with a 5-minute warm-up consisting of marching on the spot, gentle range-of-motion exercises for the lower limbs, trunk rotations, and breathing exercises. Balance training for 15 minutes will include anticipatory control exercises (such as sit-to-stand variations, weight-shifting, and stepping strategies), reactive postural control using gentle multidirectional perturbations and stepping practice, and sensory strategies like tasks on foam or uneven surfaces with eyes closed. Progression will be achieved by narrowing the base of support and adding dual-task activities. Gait training for 10 minutes will include overground walking with a focus on step length, cadence, turns, and obstacle negotiation, combined with cueing strategies such as a metronome or visual tape markers. Strengthening and core exercises for 7-10 minutes will include
  Interventions: Behavioral: Virtual Reality-Based Physical Therapy

INTERVENTIONS:
Behavioral: Conventional Physical Therapy — ntervention Description - Conventional Physical Therapy
  Conventional physical therapy consists of therapist-guided exercises aimed at improving balance, gait, strength, and functional mobility in individuals with Parkinson's disease. Each session includes a warm-up, structured balance training (anticipatory, reactive, and sensory strategies), overground gait training with cueing techniques, lower-limb and core strengthening exercises, and a cool-down period with stretching and fall-prevention education. Treatment is delivered by licensed physiotherapists three times per week for eight weeks, with exercise difficulty progressively adjusted according to individual performance and tolerance.
  Arms: group A Conventional physical therapy
Behavioral: Virtual Reality-Based Physical Therapy — Intervention Description - Virtual Reality-Based Physical Therapy
  Virtual reality-based physical therapy uses interactive computer-generated environments to provide task-specific balance and gait training with real-time visual and auditory feedback. Participants perform activities such as weight shifting, stepping to virtual targets, obstacle negotiation, and dynamic walking tasks designed to challenge postural control and mobility. Sessions are supervised by trained physiotherapists and delivered three times per week for eight weeks. Task difficulty is progressively increased based on participant performance, with safety measures in place throughout the intervention.
  Arms: group B Virtual Reality-Based Physical Therapy

SUMMARY:
Parkinson's disease is a long-term neurological condition that affects movement, balance, and daily activities. People with Parkinson's disease often experience symptoms such as slowness of movement, stiffness, tremors, and difficulty with walking and balance. Physical therapy is commonly used to help improve mobility and quality of life in these patients.

This study aims to compare virtual reality-based physical therapy with conventional physical therapy in individuals diagnosed with Parkinson's disease. Virtual reality therapy uses interactive computer-based exercises, while conventional physical therapy includes traditional exercises provided by a physiotherapist.

Participants will be randomly assigned to one of two groups. One group will receive virtual reality-based physical therapy, and the other group will receive conventional physical therapy. Both groups will follow structured treatment programs over a defined period. Outcomes such as balance, mobility, walking ability, and functional independence will be assessed before and after the intervention.

The results of this study may help determine whether virtual reality-based physical therapy is more effective, equally effective, or less effective than conventional physical therapy for improving movement and daily functioning in people with Parkinson's disease.

DETAILED DESCRIPTION:
This study is a randomized controlled trial designed to compare the effects of virtual reality-based physical therapy and conventional physical therapy on balance, gait, and fall risk in individuals with Parkinson's disease. The trial will be conducted at Shadman Medical Centre and will follow a parallel-group design. The total duration of the study will be approximately nine months following approval of the research synopsis, which will include participant recruitment, intervention delivery, follow-up assessments, and data analysis.

A total of 62 participants will be enrolled, accounting for an anticipated attrition rate of 20%. The sample size was calculated to detect clinically meaningful differences between groups with 80% statistical power at a 95% confidence level. Participants will be adults aged 45-65 years with a confirmed diagnosis of Parkinson's disease and sufficient cognitive capacity to understand instructions and participate safely in the intervention. Both male and female participants will be included. Individuals with other neurological disorders, recent musculoskeletal trauma or surgery affecting mobility or balance, or conditions that significantly impair safe participation will not be enrolled.

Participants will be recruited using a convenience sampling method and will undergo baseline assessment prior to group allocation. Randomization will be carried out using a lottery method, with allocation occurring after baseline measurements. Outcome assessors and data analysts will remain blinded to group assignment in order to minimize assessment and analysis bias.

Participants will be allocated to either conventional physical therapy or virtual reality-based physical therapy. All interventions will be delivered by licensed physiotherapists who are trained in the standardized study protocol. Both groups will receive three treatment sessions per week for eight weeks, resulting in a total of 24 sessions. Each session will last approximately 45 minutes, including warm-up and cool-down periods. Exercise intensity will be maintained at a moderate level and monitored using the Borg CR10 scale. Participants will continue their stable anti-parkinsonian medication regimen throughout the study period.

Standard safety measures will be implemented for all participants, including pre-session screening of vital signs, continuous therapist supervision, fall-risk monitoring, and use of gait belts when required. Attendance will be documented for each session, and adherence to the intervention will be defined as completion of at least 80% of the prescribed sessions.

Conventional physical therapy will focus on improving balance, gait, strength, and functional mobility through structured exercise sessions. The intervention will include balance training targeting anticipatory, reactive, and sensory integration strategies, gait training with cueing techniques, strengthening of lower-limb and core musculature, and stretching exercises during the cool-down phase. Exercise difficulty and progression will be individualized based on participant performance and tolerance.

Virtual reality-based physical therapy will involve interactive balance and gait training using immersive or semi-immersive virtual environments. Participants will engage in task-oriented activities such as weight shifting, stepping to visual targets, dynamic balance challenges, and gait-related tasks enhanced by real-time visual and auditory feedback. Reactive balance training and dual-task components may be incorporated to simulate functional and environmental demands. Task difficulty will be progressively adjusted according to performance-based criteria, with therapist supervision to ensure safety.

Outcome assessments will be conducted at baseline, mid-intervention, and post-intervention using standardized and validated clinical assessment tools administered by trained assessors in a controlled clinical environment. Assessment procedures will be standardized across all time points to ensure consistency and reliability of measurements.

Ethical approval for the study has been obtained from the Institutional Review Board of the University of Lahore. Written informed consent will be obtained from all participants prior to enrollment. Participant confidentiality will be strictly maintained through anonymization and secure handling of data. Participation will be voluntary, and participants may withdraw from the study at any time without penalty or effect on their standard medical care. All potential risks and benefits will be explained in advance, and participant safety will remain a priority throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Parkinson's disease. Patients with good cognitive status(MMSE 24 and above) Patients age range from 45- 65 Both male and female population included.

Exclusion Criteria:

* Other neurological conditions e.g. stroke, multiple sclerosis. Patients with fracture of lower limb in previous 6 months. Patients with recent major surgery or trauma of peripheries that affect mobility and balance.

Patient with spinal cord injury.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-18 (Estimated)

PRIMARY OUTCOMES:
Balance and Mobility | Baseline, (2 weeks)then (4 weeks)
  Description: Functional mobility and dynamic balance measured by the Timed Up and Go (TUG) test, which assesses the time it takes a patient to stand up from a chair, walk 3 meters, turn, walk back, and sit down.

SECONDARY OUTCOMES:
Fall Risk | Baseline, (2 weeks)then (4 weeks)
  Assessed using the Fall Efficacy Scale-International (FES-I), which evaluates fear of falling and confidence in performing daily activities without falling.

CONTACTS AND LOCATIONS:
Overall Officials: Montiha Azeem, MSPTN, Principal Investigator — The University of Lahore, Lahore
Locations (1):
- Shadman Medical Center, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No